CLINICAL TRIAL: NCT06661122
Title: An Observational Study of Darolutamide in Addition to Standard Androgen Deprivation Therapy and Docetaxel in Patients With Low-volume Metastatic Hormone-sensitive Prostate Cancer
Brief Title: A Study to Learn About How Safe Darolutamide is and How Well it Works in Combination With Androgen Deprivation Therapy and Docetaxel in Routine Medical Care for Japanese Men With Low Volume Metastatic Hormone-Sensitive Prostate Cancer
Acronym: HAYATE
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22842
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer (mHSPC); Low-volume Metastasis
Keywords: mHSPC
MeSH Terms: interventions — darolutamide; Docetaxel; Androgen Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mHSPC patients: Adult male patients with a diagnosis of low-volume metastasis HSPC (hormone-sensitive prostate cancer) whom the decision for treatment with darolutamide in combination with docetaxel and ADT has been made by the physician or a delegate.
  Interventions: Drug: Darolutamide (BAY1841788) + docetaxel + ADT

INTERVENTIONS:
Drug: Darolutamide (BAY1841788) + docetaxel + ADT — Follow clinical practice/administration. ADT=androgen deprivation therapy.

SUMMARY:
This is an observational study in which medical records of Japanese men with low-volume metastatic hormone-sensitive prostate cancer (mHSPC), who received treatment with a combination therapy of darolutamide with an androgen deprivation therapy (ADT) and docetaxel, will be collected and studied.

The study drug darolutamide, in combination with ADT and docetaxel is an approved treatment for another type of prostate cancer. To better understand the impact of this combination therapy on low-volume mHSPC and make better treatment choices, more knowledge is needed. ADT is a hormone therapy that lowers the level of testosterone, a male hormone, and slows down the growth of cancer cells. Darolutamide blocks androgen signals to slow the growth of the cancer cells. Docetaxel is a type of chemotherapy used to treat different types of cancer. It works by stopping the growth and spread of cancer cells.

The prostate gland is a male reproductive gland found below the bladder. Low-volume mHSPC is a cancer of the prostate gland that has spread beyond the gland to three or fewer bones but has not reached organs like the lungs and liver. The prostate cancer is considered hormone sensitive when it responds to an anti hormonal therapy.

In this study, only observations from routine clinical practices will be made. Participants will receive darolutamide, in combination with ADT and docetaxel as prescribed by their doctors during routine medical care. The participants will not receive any advice on treatment or any changes to healthcare as a part of the study.

The main purpose of this study is to learn more about how safe darolutamide is and how well it works in combination with ADT and docetaxel in adult Japanese men with mHSPC in routine medical care.

To do this, researchers will assess the following information about participants after one year of receiving the combination therapy by their doctors:

• the number of participants who achieve normal levels of prostate specific antigen (PSA).

PSA is a protein found in the blood that helps doctors monitor prostate cancer.

• the number of participants who have adverse events (AEs), serious adverse events (SAEs), and adverse events of special Interest (AESIs) that lead to discontinuation or change in the dose of darolutamide or docetaxel during the study.

AEs are medical problems that the participants had during the study that may or may not be related to the study treatment.

SAEs are AEs that lead to death, puts the participant's life at risk, requires hospitalization, causes disability, causes a baby to be born with medical problems, or is medically important.

AESIs are specific medical problems the participants had during the study that may be related to heart, lung, liver etc.

The data will come from the participant's medical records and will be collected between October 2024 and June 2031. Researchers will only look at the health records from adult men with mHSPC in Japan. No separate visits are required as part of the study. The participants will only visit their doctor at the study clinic as part of their routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of prostate.
* Patients have low-volume of metastatic disease documented by either by a positive bone scan, or for soft tissue either by contrast-enhanced abdominal/pelvic/chest computed tomography (CT) or magnetic resonance imaging (MRI) scan assessed by investigator. Low-volume metastasis criteria is defined as "not" meeting the high-volume criteria of the CHAARTED trial; high-volume meet the presence of visceral metastases, or four or more bone lesions including at least one outside the vertebral column or pelvis.
* Documented diagnosis of mHSPC.
* Patients on triplet regimen previously decided by the investigator irrespective of enrollment in the study.
* Start ADT within 6 months before or at the index date.
* Signed informed consent: If an eligible patient is deceased at the time of study initiation, informed consent from the legally representative(s) of the patient is required. Opt-out consent is acceptable in accordance with the Ethical Guidelines for Medical and Health Research Involving Human Subjects only when it is difficult to obtain signed informed consent from the patient or their legal representative.

Exclusion Criteria:

* Patients treated with docetaxel before darolutamide start.
* Participation in an investigational program with interventions outside of routine clinical practice.
* Contra-indications to darolutamide, docetaxel and ADT according to the local marketing authorization.
* Participation in the PASS of darolutamide in patients with mHSPC (DADOX [NCT06010914]).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients over the age of 18 years with a diagnosis of low-volume metastasis HSPC whom the decision for treatment with darolutamide in combination with docetaxel and ADT has been made by the physician or a delegate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with absolute prostate-specific antigen (PSA) response at 12 months | after 12 months
  Absolute PSA response is defined as blood PSA level <0.2 ng/mL during treatment period. Proportion of patients with absolute PSA response is defined as the number of patients with absolute PSA response, divided by the total number of patients evaluable for absolute PSA response. Proportion of patients with absolute PSA response will be evaluated on patient data up to 12 months after index date.
Number of patients with adverse event of special interests (AESIs), serious adverse events (SAEs) and adverse events (AEs) leading to dose modification or discontinuation of darolutamide or docetaxel at 12 months | after 12 months
  AESIs are defined as: Cardiac disease, Interstitial lung disease, Liver dysfunction, Neutropenia, Febrile neutropenia, Thrombocytopenia, Hypertension, Anemia, Hyperglycemia, Urinary tract infection, Decreased appetite, Fatigue, Nausea, Peripheral neuropathy, Dysgeusia.

SECONDARY OUTCOMES:
Real-world time to PSA progression in patients who have a documentation of PSA | up to 12 months
  PSA progression is defined as a ≥ 25% PSA increase above the nadir value and an increase in absolute value of ≥2 ng/mL above nadir. The time to PSA progression is defined as the time from index date to the date of first PSA progression.
Real-world time to castration-resistant prostate cancer (CRPC) | up to 12 months
Time to initiation of subsequent systemic antineoplastic therapy | up to 12 months
Time to first symptomatic skeletal event (SSE) | up to 12 months
  An SSE is defined as external beam radiation therapy (EBRT) to relieve skeletal symptoms, or new symptomatic pathologic bone fracture, or occurrence of spinal cord compression or tumor-related orthopedic surgical intervention, whichever comes first.
Time to initiation of opioid use for ≥7 consecutive days in patients who are opioid-free at baseline | up to 12 months
Dosing patterns of darolutamide and docetaxel up to 12 months | after 12 months
  The darolutamide and docetaxel administration patterns will be summarized as dosage (initial, overall), duration of administration, number of cycles administered (docetaxel only), dose modification, relative dose intensity (RDI), reason of dose modification or discontinuation.
Summary description of patient demographics / characteristics | after 12 months
  Age at baseline, Age category, Race (Japanese or not), Physical examination including height and weight, Body Mass Index (BMI), BMI category, Comorbidities (Cardiac disease, Lung disease, Liver dysfunction, etc.), ECOG PS (Eastern Cooperative Oncology Group Performance Status), and other medical history.
Summary description of laboratory values | after 12 months
  Descriptive statistics (i.e. number of observations) will be presented for the laboratory values, their changes from baseline (including baseline value), and their percent changes from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.